CLINICAL TRIAL: NCT03554200
Title: Effect of Empagliflozin on Cardiac Output in Patients With Acute Heart Failure (EMPA Acute Heart Failure)
Brief Title: EMPA Acute Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID 19
Sponsor: RWTH Aachen University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-156; 2017-002695-45 (EudraCT Number)
Record Dates: First submitted 2018-05-17; First posted 2018-06-13 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 2; Acute Heart Failure
Keywords: Empagliflozin; acute heart failure; cardiac output; left ventricular systolic and diastolic function; exercise capacity
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Single center, prospective, placebo-controlled, double blind, randomized, 2-arm parallel, interventional, exploratory pilot study
Who Masked: Participant, Investigator
Masking Description: This trial is double-blinded. After randomization neither the patients nor the investigator will be aware of the treatment allocation. Patients assigned to one of the double-blinded treatment will take one tablet Empagliflozin or matching placebo. The tablets will be identical in appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Experimental): Patients will receive empagliflozin 10 mg qd for a period of 30 days.
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Patients of the placebo arm will receive placebo tablets qd for a period of 30 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Standard of Care + Empagliflozin: 10 mg (tablets) once daily
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo — Standard of Care + Placebo: Matching Placebo (tablets) once daily
  Arms: Placebo

SUMMARY:
In this study the investigators are aiming to treat patients with acute heart failure with or without diabetes with Empagliflozin or placebo. Given the beneficial effects of Empagliflozin on heart failure hospitalization in the EMPA-REG OUTCOME trial, the investigators do expect a similar beneficial effect to be present in patients with acute heart failure. Acute heart failure is a state of hydropic decompensation resulting in dyspnea and congestions, caused by different etiologies of cardiac disease. Recompensation is reached by application of diuretic drugs and fluid restriction.

DETAILED DESCRIPTION:
In the present study patients will be randomized into 2 groups (standard of care + Empagliflozin 10 mg/d or standard of care + placebo). Cardiac output will be assessed by a medical device for noninvasive monitoring of hemodynamic parameters (cardiac output, systemic vascular resistance, stroke volume and blood pressure) using finger cuff technology for pulse contour analysis.

These investigations will inform about Empagliflozin dependent effects on hemodynamic and cardiac function in patients with acute heart failure. The investigation will further assess the therapeutic efficacy of Empagliflozin on heart failure symptoms using objective (respiratory rate, oxygen requirement, peak expiratory flow rate, urinary volume, body weight, diuretic requirement, length of hospital stay) and well accepted, patient orientated secondary endpoints. In addition, metabolic regulators and parameters relevant for cardiac function and substrate metabolism will be assessed to further investigate possible mechanisms of Empagliflozin-dependent actions on cardiac function.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with acute heart failure with associated signs or symptoms (dyspnea on exertion, orthopnea, paroxysmal dyspnea, peripheral oedema, chest x-ray with pulmonary congestion)
3. Serum levels of NT-proBNP ≥ 1000 pg/ml within 48 hours of Informed Consent
4. Written informed consent prior to study participation

Exclusion Criteria:

1. Type 1 diabetes
2. Participants of child-bearing age without adequate contraception
3. Pregnancy or lactating females
4. Cardiogenic shock
5. Acute coronary syndrome within 30 days prior to randomization
6. Planned or recent percutaneous or surgical coronary intervention within 30 days prior to randomization
7. Signs of ketoacidosis and/or hyperosmolar hyperglycemic syndrome (pH ≤ 7.30 and glucose >14 mmol/l and HCO3- ≤ 18 mmol/l)
8. Signs of uncontrolled active infection
9. Dyspnea due to non-cardiac causes (severe pulmonary disease, anemia, severe obesity), non-HF causes such as acute or chronic respiratory disorders
10. Coronary artery disease with requirement for revascularization within the study period
11. Renal impairment (GFR < 20 ml/min/1,73 m2)
12. Known hepatic impairment (as evidenced by total bilirubin >3 mg/dL) or history of cirrhosis with evidence of portal hypertension (e.g., presence of esophageal varices)
13. Uncontrolled thyroid disease
14. Endocrinopathies like Graves' disease, acromegaly, Cushings' disease
15. Hypertensive retinopathy or encephalopathy
16. Bariatric surgery in last 2 years prior to randomization
17. Patients in whom study participation is not deemed appropriate under consideration of clinical wellbeing by the principal investigator
18. The subject is mentally or legally incapacitated
19. The subject received an investigational drug within 30 days prior to inclusion into this study
20. Urinary tract infections or significant formation of residual urine in medical history
21. Patients with particular risk for ketoacidosis (alcohol abuse, pancreatitis, pancreatic insulin deficiency from any cause, caloric restriction etc.) or ketoacidosis in the past
22. Frequent hypoglycaemic events (in the opinion of the investigator)
23. Intolerance to Empagliflozin and excipients in Empagliflozin or rather placebo
24. Patients with severe stenosis or regurgitation of the aortic, pulmonary or mitral valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
effect of Empagliflozin 10mg qd versus placebo on cardiac output in patients with acute heart failure | 30 days
  by ClearSight System

SECONDARY OUTCOMES:
Hemodynamics | 30 days
  Systemic vascular resistance (mmHg⋅min⋅mL-1)
Hemodynamics | 30 days
  Stroke volume (ml/beat)
Exercise Capacity | 30 days
  Hand grip
Cardio vascular | 30 days
  blood pressure (mmHg)
Effect of Empagliflozin on systemic quality of life | 30 days
  Quality of life questionnaire
Effect of Empagliflozin on hospitalization due to cardiovascular causes or readmission for heart failure or renal failure | 30 days
  length of initial hospital stay
Effect of Empagliflozin on death due to cardiovascular causes | 30 days
  days alive and out of hospital
Urine | 30 days
  24 h sodium excretion (mmol/day)
Body weight | 30 days
  body weight (kg)
Cardio vascular | 30 days
  24 h heart rate (bpm)
Blood | 30 days
  NT-proBNP (ng/l)
Blood | 30 days
  cystatin C(mg/dl)
Blood | 30 days
  serum levels of Glucose, Glucagon, Insulin, Total-Ketone bodies, Hydroxybutyrate, Aldosterone, Free fatty acidy (mg/dl)
Blood | 30 days
  Hemoglobin, Haematocrit, Erythropoietin
Respiratory rate | 30 days
  breaths/min
Diuretic response | 30 days
  Δ weight kg/[(total i.v. dose)/40mg]+[(total oral dose)/80mg)] furosemide
Kidney injury risk score | 30 days
  by NephroCheck® (defined by TIMP-2 x IGFBP7 in urine)
change of microbiome | 30 days
  stool sample
Patient-reported dyspnea | 30 days
  visual analogue scale (VAS), 7 point categorical Likert scale
Peak expiratory flow rate | 30 days
Oxygen | 30 days
  Saturation (%)
Oxygen | 30 days
  delivered (l/min)
Clinical judged diuretic requirement | 30 days
Blood | 30 days
  eGFR
Blood | 30 days
  Lactate, pH, HCO3-
Blood | 30 days
  Serum osmolarity, Potassium, Chloride
Effect of Empagliflozin 10 mg daily on Left ventricular systolic function | 30 days
  ejection fraction
Effect of Empagliflozin 10 mg daily on Left ventricular diastolic function | 30 days
  2D and 3D parameter global strain rate E by echocardiography and by standardized parameter E/E' and left atrial (LA) volume

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine I RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No